CLINICAL TRIAL: NCT01620268
Title: An Open-Label, Phase 2 Study to Treat Patients With Renal Allograft and Polyoma BK Viruria to Prevent Polyoma BK Viremia, Polyoma BK Nephropathy and Renal Allograft Rejection
Brief Title: An Open-Label, Study to Treat Patients With Renal Allograft and Polyoma BK Viruria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Changzheng-Cinkate (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CK2012-001
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Viruria; Viremia
Keywords: leflunomide; orotic acid; Polyoma BK Viruria; Polyoma BK Viremia; Polyoma BK Nephropathy; Renal Allograft Rejection
MeSH Terms: conditions — Viremia | interventions — Leflunomide; Orotic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Patients receive standard of care.
- Treatment Group (Experimental): Dose adjusted leflunomide plus 600 mg orotic acid.
  Interventions: Drug: Leflunomide and orotic acid

INTERVENTIONS:
Drug: Leflunomide and orotic acid — Daily dose of leflunomide adjusted to target steady state blood levels of 50 ug/mL to 100 ug/mL of the active metabolite plus 600 mg orotic acid
  Arms: Treatment Group

SUMMARY:
This study will evaluate the clinical efficacy and safety of a combination of leflunomide and orotic acid in kidney transplant patients with high levels of Polyoma BK viruria for the purpose of preventing Polyoma BK viremia and Nephropathy that could lead to kidney transplant loss from viral damage, acute rejection or both.

DETAILED DESCRIPTION:
This is a multicenter, randomized trial that will evaluate the effect of a combination of leflunomide and orotic acid for the treatment of Polyoma BK viruria. In this multicenter trial, renal allograft patients with the diagnosis of Polyoma BK viruria as determined by a viral level in the urine of 25 million or more copies/mL, and no detectable viremia, will complete a screening visit (V1) to determine eligibility for the study based on inclusion/exclusion criteria. Patients that meet the entrance criteria for this study will be randomly assigned to one of two treatment groups at Visit (2) and enter a 4 month dosing period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, 75 years of age or less, with the diagnosis of renal allograft Polyoma BK viruria of 10 million or more copies/mL in their urine confirmed by PCR at the central laboratory.
2. No viremia (viremia is defined as greater than 1,000 copies/ml plasma on two consecutive tests two weeks or more apart as measured at the designated central laboratory),
3. Serum creatinine <2.0 mg/dL
4. Hct > 30%
5. WBC > 3,500 x 103/L
6. Platelet count > 150,000 x 103/L
7. Normal values for ALT, AST and bilirubin; Alk Phos < 2 X upper limits of normal
8. No symptomatic cardiac, pulmonary, GI, hepatic or neurologic disease
9. No other active infections
10. Receiving CyA or Tacrolimus, Mycophenolate/Azathioprine + prednisone.
11. Is not pregnant as verified by a pregnancy test

Exclusion Criteria:

1. Is not able to comply with study procedures and dosing.
2. Has psychiatric instability.
3. Has an active systemic infection including Hepatitis B or C, HIV, or on anti-viral therapy within seven days of entering the study. Note however, that the subjects may be taking ganciclovir, valaciclovir, acyclovir and valganciclovir and therefore these are not exclusionary antiviral medications.
4. Has BK viremia (viremia is defined as greater than 1,000 copies/ml plasma on two consecutive tests two weeks or more apart as measured at the designated central laboratory), or has had a single episode of BK viremia. (viremia is defined as greater than 1,000 copies/ml plasma on two consecutive tests two weeks or more apart as measured at the designated central laboratory or the local laboratory),
5. Has a cancer diagnosis within past five years with potential for recurrence.
6. Has received experimental drug within past 3 months.
7. Is receiving immune suppressive drug other than those listed above calcineurin inhibitor, mycophenolate/azathioprine and +/- corticosteroid)
8. Is a woman of child bearing potential or is a male with female partner of child bearing potential who is unwilling to use reliable contraception.
9. Has any neurologic abnormalities including peripheral neuropathy.
10. Is receiving concomitant therapy with drug known to have hepatotoxic risk.
11. Has known or suspected liver disease or current alcohol abuse.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Clearance of viruria | 12 weeks
  Viral load of Polyoma BK virus in urine reduced from greater than or equal to 10 million copies/mL to less than 500,000 copies/mL or a 2 log reduction in copies/mL.

SECONDARY OUTCOMES:
Absence of viremia | 12 weeks
  No more that 1000 copies of Polyoma BK Virus in the blood on two consecutive tests 2 weeks or more apart
Absence of Polyoma BK Nephropathy | 12 weeks
  Absence of Polyoma BK Nephropathy
No rejection of the renal allograft | 12 weeks
  No rejection of the renal allograft

CONTACTS AND LOCATIONS:
Overall Officials: James W Williams, MD, Principal Investigator — Cinkate Corp
Locations (9):
- United States (9):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Tampa General Hospital, Tampa, Florida
  - Rush Univeristy, Chicago, Illinois
  - University of Illinois, Chicago, Chicago, Illinois
  - The University of Chicago Transplant Center, Chicago, Illinois
  - IU Health, Indianapolis, Indiana
  - University of Lousiville, Louisville, Kentucky
  - Beth Israel Deaconess Hospital, Boston, Massachusetts
  - Methodist University Hospital, Memphis, Tennessee